CLINICAL TRIAL: NCT06973460
Title: Investigating the Role of a Robotic-Assisted System in Enhancing Balance, Postural Stability, Functional Gait and Fall Efficacy in Older Adults Compared to Balance and Mobility Exercise - A Pilot Study
Brief Title: Robotic-Assisted System in Enhancing Balance, Postural Stability, Functional Gait and Fall Efficacy in Older Adults
Acronym: ROB-BST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gulf Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB-COHS-STD-96-Nov-2024
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Aged; Aged Healthy Volunteer; Geriatric; Balance; Fall Risk, Fall Prevention
Keywords: Robotic System; Hunova; Balance; Older Adults; Fall Efficacy; Functional Gait; Robotic-assisted System; Balance and Mobility Exercise; Otago Exercise Programme

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Robotic Assisted Group Using the Hunova Movendo Robotic Device. (Experimental): Balance Training on Robotic Assisted System:
  Bipodalic Stance: On Static platform; Elastic Platform, Fluid platform, Wobble Base, Balance on variable counter resistance platform, Sagittal Lunges.
  Monopodalic (Left & Right): On Static platform; Elastic Platform, Fluid platform, Wobble Base, Balance on variable counter resistance platform, Isometric Ankle.
  Strengthening: Balance on Counter-resistance platform, raises, Ping Pong on Elastic platform, Bipodalic Sit to Stand
  Mobility and Gait: Bipodalic Stance: Balance on Elastic Platform, Balance on Fluid Platform, Balance on Proprioceptive Platform, Balance on Linear PAssive
  Combined Passive platform, Balance on Passive Spiral Base.
  In addition: Stair walking on standardized stairs.
  Rest Period: 5 mins incorporated in between intervention. Duration : 45 minutes/day
  Frequency:
  2 days per week for a period of 12 weeks
  Interventions: Device: Hunova Robotic-Assisted System
- Balance and Mobility Exercises derived from Otago Exercise Programme. (Active Comparator): * Strengthening Training:
  * Knee Extensor
  * Knee Flexor
  * Hip Adductor
  * Ankle plantarflexors (calf Raises)
  * Ankle dorsiflexors (toe raises)
  * Balance Training:
  * Knee Bends
  * Backwards walking
  * Walking and turning around
  * Sideways walking
  * Tandem Stance (heel toe stand)
  * Tandem Walk (Heel toe Walk)
  * One Leg Stand
  * Heel walking
  * Toe Walk
  * Heel Toe Walking backwards
  * Sit to Stand
  * Stair walking
  Rest Period: 5mins incorporated in-between intervention. Duration : 45 minutes/day
  Frequency:
  2 days per week for a period of 12 weeks
  Interventions: Other: Balance and Mobility Exercise

INTERVENTIONS:
Device: Hunova Robotic-Assisted System — Hunova Movendo Robotic System
  Arms: Robotic Assisted Group Using the Hunova Movendo Robotic Device.
Other: Balance and Mobility Exercise — Balance and Mobility Exercise derived from the Otago Exercise Programme
  Arms: Balance and Mobility Exercises derived from Otago Exercise Programme.

SUMMARY:
Our study aims to investigate the effectiveness of a more individualized and personalized feedback-oriented approach using the Hunova Robotic Systems. This system is tailored to specific needs of individuals and is dynamically adjustable relative to patients' balance and functional demands. It will be compared to Traditional Balance and Mobility Exercise which are more generalized. Given the generalized nature of Traditional approaches, we aim to compare it with the Hunova Robotic Systems in the enhancement of Balance, Postural Stability, Functional Gait and Fall Efficacy in older adults.

DETAILED DESCRIPTION:
Aging comes with increased risk of fall and a steep decline in adequate motor functioning, as such due to the decline in proprioception, balance and general functional independence the risk of falls and injury is high in aging adults impacting quality of life.

Traditional approaches like the Otago Exercise Programmes (and other Balance and Mobility exercise protocols) have been relatively effective in the management of falls yet there's a remarkable and persistent increase in fall rates, postural instability and functional gait limitations in older adults largely due to the generalized nature of these protocols. The limitations of these traditional approaches in individualizing treatment protocols created a need for advanced and more dynamic systems that can fill this gap and/or complement these traditional approaches.

Modern Technology, including Hunova Robotic systems are novel approaches that seek to solve these limitations by tailoring interventions to patients' needs creating real time feedback mechanisms assisting in intervention prescriptions and analysis. The preciseness of these modern systems assist in creating integrated systems that enhance organization of these interventions improving overall outcomes.

Literature supporting the use of the Hunova Robotic System on Fall efficacy, postural stability and functional gait is very limited, necessitating a need for studies comparing the effectiveness of this technology on these components compared to Traditional Balance and Mobility Exercise Protocols. This research aims to investigate the effectiveness of Movendo's Hunova in improving fall efficacy, postural stability and functional gait in older adults and in general geriatric rehabilitation. With the increased emphasis on robotic-assisted rehabilitation due to its accuracy, individualized patient focused design and feedback mechanisms, the study becomes all the more imperative.

This Research attempts to compare the Hunova Robotic System on Fall Efficacy, Functional Gait and postural stability with traditional balance and Mobility Exercise Protocols.

ELIGIBILITY:
Inclusion Criteria:

* 60 years old to 85 years old - young to Old Individuals.
* Mini Mental Scale Examination Score > 24.
* Able to walk independently with and without mild assistance (Berg's Balance Score between 35 and 45)

Exclusion Criteria:

* Unable to understand and follow instructions.
* History of vestibular dysfunction.
* Any severe Musculoskeletal problems restricting mobility.
* Current Physiotherapy training or balance exercises focusing on proprioception or fall risk.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Hunova Evaluation Tools: | Baseline and 12 weeks
  Hunova's precise assessment tools assist clinicians tailor prevention interventions with Quantitative data.
  Assessment Domains:
  Static & dynamic postural control Visual dependency in balance (Romberg Index) Trunk stability Functional sit-to-stand transitions Limits of stability
  Scoring:
  No single cumulative score; results are reported through individual biomechanical parameters such as:
  Sway Area (cm²) (CE,OE) COP Path Length (cm) (CE,OE) Romberg Index (unitless ratio) Trunk Oscillation Range (deg) (multi directionally) (CE,OE) 5x Sit-to-Stand Duration (seconds) Limits of Stability (LoS) (cm) (Max COP & LEAN multi directionally).
  Interpretation:
  Lower values (individualized normative values) in Sway Area, Path Length, & Romberg Index indicate better balance, greater postural control, & lower fall risk.
  Higher values (individualized normative values) in Trunk Oscillation, LoS & Sit-to-Stand times reflect reduced functional stability & potential impairments in dynamic control.

SECONDARY OUTCOMES:
Berg's Balance Scale (BBS) | Baseline and 12 weeks
  A Gold Standard in the assessment of Balance Impairments
  Score range: 0 to 56
  Interpretation: Higher scores indicate better balance and lower fall risk.
Star Excursion Balance Test (SEBT) | Baseline and 12 weeks
  This test assesses dynamic balance by measuring reach distance while balancing on one leg in various directions. Used to detect deficits in balance and flexibility, it has an interrater reliability and has been validated in the identification of balance deficits in lower extremity. It is useful in assessment of the functional strength of older adults as they're prone to balance, proprioception and flexibility decline.
  Range: Reach distance measured in centimeters; often normalized to leg length.
  Intepretation: Greater reach distance indicates better dynamic postural control.
Functional Gait Assessment (FGA): | Baseline and 12 weeks
  FGA is an assessment scoring scale that measures gait stability under different conditions and tasks. It ranges from 0-30. Lower scores signify higher gait impairments. It has an interrater reliability (ICC > 0.9). It also has high sensitivity to functional gait changes supporting its use care in baseline and follow up assessments in Older Adults
Fall Efficacy Scale- International (FES-I): | Baseline and 12 weeks
  FES-I is a 16 to 64 self-reporting tool that is used to assess confidence in performing activities without the risk of fall. Higher scores signify a greater fear of falling. It gives insight on how much the fear of falling influences activities. It has an internal consistency (Cronbach's Alpha > 0.9) suggesting reliability and validity in research

CONTACTS AND LOCATIONS:
Overall Officials: Meruna Bose, PHD, Study Chair — Gulf Medical University
Locations (1):
- Thumbay Physical Therapy and Rehabilitation Hospital, Ajman, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No
Data might be shared based on the request